CLINICAL TRIAL: NCT05413317
Title: Contribution of Lower Limb Venous Colour Doppler Ultrasound in the Diagnosis of Pulmonary Embolism Recurrence
Acronym: RECHOPE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-CHITS-012
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary embolism; Deep vein thrombosis; Recurrence; Diagnosis strategy; Colour Doppler ultrasound
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients hospitalized for suspicion of pulmonary embolism recurrence: Patients with at least one of the following symptoms: acute dyspnea or aggravation of chronic dyspnea, chest pain, hemoptysis or syncope
  Interventions: Other: Color Doppler Ultrasound

INTERVENTIONS:
Other: Color Doppler Ultrasound — Comparison with conventional diagnosis strategy including a clinical probability score, D-dimers and chest imaging.
  Other Names: Diagnosis strategy

SUMMARY:
Venous thromboembolic disease is a clinical entity including pulmonary embolism (PE) and deep vein thrombosis (DVT). It is a chronic disease with 30% recurrence rate at 10 years. In patients with recurrent PE clinical suspicion, an objective and accurate diagnostic method/strategy is warranted to exclude or confirm a PE new episode diagnosis and to decide on treatment initiation.

Recurrent PE diagnosis raises several issues related to the limitations of clinical scores, D-dimer testing, and diagnostic imaging used for a first episode diagnosis. Most importantly, residual obstruction on chest imaging reported in more than 50% of cases at 6 months can make it difficult to distinguish between an old and a new thrombosis in the absence of possible comparison with a previous imaging carried out under the same modalities.

There are currently few recommendations about the diagnostic strategy for patients with a recurrent PE clinical suspicion and these recommendations are not very consistent due to the lack of a validated strategy. None of current guidelines have included imaging-detectable lower-limb DVT within the strategies despite a reported high prevalence of PE-associated DVT. In one study using venography, 82% (95% CI 76.5 - 86.9) of angiographically-proven PE patients had an associated proximal or distal deep vein thrombosis, of which 42% were asymptomatic. In another study using lower-limb venous ultrasound, a proximal or distal DVT was detected in 93% (95% CI 85-97) of patients with PE.

DETAILED DESCRIPTION:
In this study, patients with PE clinical suspicion and a previous PE episode have a standard diagnostic work-up based on clinical probability assessment, D-dimer testing and diagnostic imaging (pulmonary CT angiography, ventilation perfusion scan).

A bilateral lower-limb venous colour doppler ultrasound (CDUS) is performed in parallel in these patients as usually carried out in our hospital for the diagnosis management of patients with clinically suspected PE. This test is performed and interpreted by an independent sonographer unaware of the results of the standard diagnostic work-up.

Lower-limb venous CDUS is then compared to the results of the standard work-up as interpreted during expert panel meetings by members involved in the diagnosis and management of patients with PE and DVT.

Data will be collected both retrospectively and prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Adult consecutive patients (>= 18 years old)
* Hospitalized for clinical suspicion of pulmonary embolism recurrence with at least one of the following symptoms: acute dyspnea or worsening of chronic dyspnea, chest pain, hemoptysis or syncope

Exclusion Criteria:

* Time between onset of symptoms and diagnosis > 15 days
* Pregnant women
* Contra-indication to CT pulmonary angiography
* Lower-limb CDUS not possible to perform for technical reasons
* Lung scans not possible to perform for technical reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized for suspicion of pulmonary embolism recurrence
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2023-11-04 (Actual); Study Completion 2023-11-04 (Actual)

PRIMARY OUTCOMES:
To evaluate lower-limb venous Color Doppler Ultrasound (CDUS) contribution to the conventional strategy used for pulmonary embolism recurrence diagnosis including a clinical probability score, D-dimers and chest imaging. | At diagnostic work-up (24 first hours following admission)
  Proportion of patients for whom the lower-limb venous CDUS is positive. CDUS will be considered as positive if an acute DVT is shown with any of the following aspects:
  * Mobile thrombus
  * Completely occlusive thrombus
  * Sub-occlusive thrombus without deep venous reflux
  Color Doppler Ultrasound will be considered as negative for a new thrombosis if the vein is compressible and there is no image of DVT, or if there are images of DVT sequelae only, with one of the following aspects:
  * Parietal residual sequelae
  * Partial obstruction with deep venous reflux

SECONDARY OUTCOMES:
To compare demographic characteristics between groups of patients with and without a new episode of PE based on expert panel decision and lower limbs CDUS results. | At diagnostic work-up (24 first hours following admission)
  Statistical analysis of the following characteristics based on demographic variables usually collected in our hospital during patient management : Age, gender, height, weight, BMI.
To compare clinical characteristics between groups of patients with and without a new episode of PE based on expert panel decision and lower limbs CDUS results. | At diagnostic work-up (24 first hours following admission)
  Statistical analysis of the following characteristics based on clinical variables usually collected in our hospital during patient management :
  * Vital signs: temperature, systolic blood pressure, diastolic blood pressure, heart rate, peripheral oxygen saturation (%)
  * Clinical scores: diagnostic (Wells score), prognostic (sPESI, ESC)
  * Symptoms: dyspnea, chest pain, malaise, hemoptysis, lower limb edema, lower limb redness, lower limb pain
  * History of venous thromboembolic disease (details)
  * Context: presence or absence of risk factors for venous thromboembolic disease
  * Comorbidities: chronic respiratory failure, chronic heart failure, hemorrhagic or ischemic stroke, hypertension, dyslipidemia, smoking, cancer
  * Treatment: antiplatelet, anticoagulant, anti-inflammatory, hormonal treatment, chemotherapy
To compare biological characteristics between groups of patients with and without a new episode of PE based on expert panel decision and lower limbs CDUS results. | At diagnostic work-up (24 first hours following admission)
  Statistical analysis of the following characteristics based on blood tests usually performed in our hospital during patient management :
  * Hemoglobin, neutrophil/lymphocyte ratio, D-dimer
  * Creatinine clearance expressed as Cockcroft and Gault (mL/min), CRP (mg/L)
  * NT-proBNP, troponin, fibrinogen
To compare imaging characteristics between groups of patients with and without a new episode of PE based on expert panel decision and lower limbs CDUS results. | At diagnostic work-up (24 first hours following admission)
  Statistical analysis of the following characteristics based on imaging tests usually performed in our hospital during patient management :
  * CT pulmonary angiography
  * Ventilation-perfusion scan
  * Venous CDUS

CONTACTS AND LOCATIONS:
Overall Officials: Marie ELIAS, MD, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (1):
- CHITS, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heit JA, Spencer FA, White RH. The epidemiology of venous thromboembolism. J Thromb Thrombolysis. 2016 Jan;41(1):3-14. doi: 10.1007/s11239-015-1311-6. PMID 26780736
- [Background] Patel P, Patel P, Bhatt M, Braun C, Begum H, Wiercioch W, Varghese J, Wooldridge D, Alturkmani H, Thomas M, Baig M, Bahaj W, Khatib R, Kehar R, Ponnapureddy R, Sethi A, Mustafa A, Lim W, Le Gal G, Bates SM, Haramati LB, Kline J, Lang E, Righini M, Kalot MA, Husainat NM, Jabiri YNA, Schunemann HJ, Mustafa RA. Systematic review and meta-analysis of test accuracy for the diagnosis of suspected pulmonary embolism. Blood Adv. 2020 Sep 22;4(18):4296-4311. doi: 10.1182/bloodadvances.2019001052. PMID 32915980
- [Background] Nijkeuter M, Hovens MM, Davidson BL, Huisman MV. Resolution of thromboemboli in patients with acute pulmonary embolism: a systematic review. Chest. 2006 Jan;129(1):192-7. doi: 10.1378/chest.129.1.192. PMID 16424432
- [Background] Meysman M, Everaert H, Vincken W. Factors determining altered perfusion after acute pulmonary embolism assessed by quantified single-photon emission computed tomography-perfusion scan. Ann Thorac Med. 2017 Jan-Mar;12(1):30-35. doi: 10.4103/1817-1737.197772. PMID 28197219
- [Background] Sanchez O, Benhamou Y, Bertoletti L, Constans J, Couturaud F, Delluc A, Elias A, Fischer AM, Frappe P, Gendron N, Girard P, Godier A, Gut-Gobert C, Laporte S, Mahe I, Mauge L, Meneveau N, Meyer G, Mismetti P, Parent F, Pernod G, Quere I, Revel MP, Roy PM, Salaun PY, Smadja DM, Sevestre MA. [Recommendations for best practice in the management of venous thromboembolic disease in adults. Long version]. Rev Mal Respir. 2021 Apr;38 Suppl 1:e1-e6. doi: 10.1016/j.rmr.2019.05.038. Epub 2019 Jul 4. No abstract available. French. PMID 31280989
- [Background] Lim W, Le Gal G, Bates SM, Righini M, Haramati LB, Lang E, Kline JA, Chasteen S, Snyder M, Patel P, Bhatt M, Patel P, Braun C, Begum H, Wiercioch W, Schunemann HJ, Mustafa RA. American Society of Hematology 2018 guidelines for management of venous thromboembolism: diagnosis of venous thromboembolism. Blood Adv. 2018 Nov 27;2(22):3226-3256. doi: 10.1182/bloodadvances.2018024828. PMID 30482764
- [Background] Ageno W, Squizzato A, Wells PS, Buller HR, Johnson G. The diagnosis of symptomatic recurrent pulmonary embolism and deep vein thrombosis: guidance from the SSC of the ISTH. J Thromb Haemost. 2013 Aug;11(8):1597-602. doi: 10.1111/jth.12301. No abstract available. PMID 23682905
- [Background] Girard P, Musset D, Parent F, Maitre S, Phlippoteau C, Simonneau G. High prevalence of detectable deep venous thrombosis in patients with acute pulmonary embolism. Chest. 1999 Oct;116(4):903-8. doi: 10.1378/chest.116.4.903. PMID 10531151
- [Background] Elias A, Colombier D, Victor G, Elias M, Arnaud C, Juchet H, Ducasse JL, Didier A, Colin C, Rousseau H, Nguyen F, Joffre F. Diagnostic performance of complete lower limb venous ultrasound in patients with clinically suspected acute pulmonary embolism. Thromb Haemost. 2004 Jan;91(1):187-95. doi: 10.1160/TH03-05-0278. PMID 14691585